CLINICAL TRIAL: NCT04339725
Title: Research Based on Gut Microbiota Metagenomics for Prevention of Chronic Liver Disease
Brief Title: Gut Microbiota Metagenomics for Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Suk, Proffesor, Chuncheon Sacred Heart Hospital
Other Study IDs: STOOL
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Liver Disease Chronic
Keywords: Liver; Fecal; Gut microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fecal DNA: Extraction fecal DNA and compare disease group to normal group
  Interventions: Other: DNA extraction

INTERVENTIONS:
Other: DNA extraction — Extraction fecal DNA and compare disease group to normal group

SUMMARY:
Gut microbiota modulation has effect on chronic liver disease

DETAILED DESCRIPTION:
Chronic liver disease has been known as a disease of the liver which lasts over a period of 6-month. It consists of inflammation, hepatitis, cirrhosis, hepatocellular carcinoma.

Gut microbiota plays an important roles in the chronic liver disease. It can suppress the progression of the liver disease by moulation gut microbiota.

The investigators are still evaluating the effect of gut microbiota on the liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 19+
* Normal : AST or ALT level < 50IU/L, BMI < 25
* Liver disease : AST or ATL level ≥ 50IU/L, BMI ≥ 25
* Patients hospitalized with chronic liver disease (viral hepatitis, alcoholic liver disease, non-alcoholic liver disease, cirrhosis, liver cancer)

Exclusion Criteria:

* Normal : AST or ATL level ≥ 50IU/L, BMI ≥ 25
* Liver disease : AST or ALT level < 50IU/L, BMI < 25
* If the patient refuses

Ages: 31 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3240 of population stool were collected. All of them are agree to provide it to investigation.
Sampling Method: Non-Probability Sample
Enrollment: 3240 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Fecal DNA | 10 years
  Compare the species and proportions of the gut microbiome
Liver enzyme | 10 years
  Compare the liver enzyme level
BMI | 10 years
  Compare the body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park IG, Yoon SJ, Won SM, Oh KK, Hyun JY, Suk KT, Lee U. Gut microbiota-based machine-learning signature for the diagnosis of alcohol-associated and metabolic dysfunction-associated steatotic liver disease. Sci Rep. 2024 Jul 12;14(1):16122. doi: 10.1038/s41598-024-60768-2. PMID 38997279
- [Derived] Ganesan R, Gupta H, Jeong JJ, Sharma SP, Won SM, Oh KK, Yoon SJ, Han SH, Yang YJ, Baik GH, Bang CS, Kim DJ, Suk KT. Characteristics of microbiome-derived metabolomics according to the progression of alcoholic liver disease. Hepatol Int. 2024 Apr;18(2):486-499. doi: 10.1007/s12072-023-10518-9. Epub 2023 Mar 31. PMID 37000389